CLINICAL TRIAL: NCT01449149
Title: Proton Radiation For Chordomas and Chondrosarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01310
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chordomas; Chondrosarcomas
Keywords: Age 18 or greater; No prior radiation
MeSH Terms: conditions — Chordoma; Chondrosarcoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton group (Experimental): Proton radiation total dose 72.00 to 79.2 Gy(RBE) in 40-44 fractions
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy

SUMMARY:
The objectives of this study are 1) To evaluate the feasibility and acute side effects of proton therapy for chordomas and chondrosarcomas and 2) To evaluate clinical outcomes and long term side effects of proton beam radiation for treatment of chordomas and chondrosarcomas.

DETAILED DESCRIPTION:
This trial will be conducted in two phases: a feasibility then a phase II trial. Once feasibility and safety are established in the first 12 pts. the phase II study will begin. Proton therapy at standard doses is not known to improve clinical outcome but will likely reduce fatigue and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of chordoma or chondrosarcoma.
* Patients must have no evidence of metastatic disease based on routine imaging (CT or MRI of the chest/abdomen/pelvis, bone scan, etc.)
* Patients must have an ECOG score equal to or less than 2.
* Age ≥ 18 years.
* Patients must be able to provide informed consent.
* Adequate bone marrow function: WBC ≥ 4000/mm3, platelets ≥ 100, 000mm3
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive , IUD, condoms or other barrier methods etc.) Hysterectomy or menopause must be clinically documented.
* Tumors arising in the skull and spine.

Exclusion Criteria:

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma)
* Patients with the following histologies are excluded: melanoma , other soft tissue or bony sarcomas, giant cell tumor aneurismal bone cyst or metastatic lesions from other histologies.
* Pregnant women.
* Actively being treated on any other therapeutic research study.
* Tumors arising outside of the CNS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Group: Proton radiation total dose 72.00 to 79.2 Gy(RBE) in 40-44 fractions
  Proton Therapy
Period: Overall Study
Arm/Group | Proton Group
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proton Group
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 54 [23 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54
Histology [Count of Participants; unit: Participants]
  Chordoma | 42
  Chondrosarcoma | 12
Lesion site [Count of Participants; unit: Participants]
  Clivus/skull base | 39
  C spine | 3
  T spine | 0
  L spine | 1
  Sacrum/coccyx | 11

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Proton RT for Chordomas and Chondrosarcomas
Description: The purpose of this study was to evaluate the feasibility and safety of dose-escalated proton beam therapy for treating chordomas and chondrosarcomas of the skull base and spine.
  The feasibility, as defined by ≥10% of patients experiencing either: unsatisfactory dosimetry, inability to complete all of his/her treatments within 10 days of estimated completion date and requiring no break >5 days, and no greater than 20% of patients experiencing ≥grade 3 toxicity from RT.
Time Frame: From enrollment to treatment completion or withdrawal, whichever occurred first, assessed up to 133 months
Population: Follow-up
Measure: Number; unit: percentage of patients did not meet this
Arm/Group | Proton Group
Number analyzed (Participants) | 54
percentage of patients did not meet this
  >10% of patients experiencing unstatisfactory dosimetry or inability to complete his/her treatments | 3.7
  20% of patients experienceing >= grade 3 toxicity | 1.9

2. Secondary Outcome: Acute Toxicities
Description: Any grade 3 or higher toxicity observed within 90 days from start of therapy.
Time Frame: With in the 90 days from tx start date
Population: Number of cases
Measure: Number; unit: Number of cases
Arm/Group | Proton Group
Number analyzed (Participants) | 54
Number of cases
  Fatigue | 37
  Radiation dermatitis | 28
  Headache | 14
  Alopecia | 9
  Insomnia | 9
  Paresthesia | 7
  Constipation | 7
  Pain | 4
  Dysphagia | 6
  Xerostomia | 4
  Diarrhea | 2
  Anorexia | 5
  Urinary (retention or incontinence) | 6
  Ataxia | 5
  Oral mucositis | 2
  Edema | 2
  Visual/blurry | 2
  Nerve palsy | 1
  Tinnitus | 1
  Dysgeusia | 5
  Cognitive disturbance | 3
  Voice alteration | 3
  Dysarthria | 1

3. Secondary Outcome: Late Toxicities
Description: Any grade 3 or higher toxicity observed later than 90 days from completion of therapy.
  Timepoints included below:
  Approx. 90 days from tx start. Follow-Up Months (approximately from completion of treatment) 3,6,9,12,15, 18, 21, 24 (approx.) Months 30, 36 (approximately from completion of treatment) Year 4 and 5 (approximately from completion of treatment)
Time Frame: Every 3 months for 3 Years from the tx start date and assessed up to 133 months
Population: Number of cases
Measure: Number; unit: Number of cases
Arm/Group | Proton Group
Number analyzed (Participants) | 54
Number of cases
  Late Fatigue | 17
  Late Headache | 8
  Late Pain | 4
  Late Loss of smell | 1
  Late Cognitive disturbance | 2
  Late Xerostomia | 1
  Late Paresthesia | 5
  Late Insomnia | 1
  Late Diarrhea | 1
  Late Neck edema | 1
  Late Dysgeusia | 2
  Late Ataxia | 5
  Late Aphasia | 1
  Late Radionecrosis of the brain | 3
  Late Anorexia | 2
  Late Dysphagia | 2
  Late Muscle weakness | 1
  Late Intranasal carotid blowout | 1
  Late Osteoradionecrosis | 1

ADVERSE EVENTS:
Time Frame: Acute and late toxicities were assessed for a time frame of over 133 months at 3-month intervals.
Arm/Group | Proton Group
All-Cause Mortality (participants affected / at risk) | 3/54
Serious Adverse Events (participants affected / at risk) | 15/54
Other Adverse Events (participants affected / at risk) | 45/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Group (N=54)
Sensory neuropathy (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Optic nerve disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Anorectal infection (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Group (N=54)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 5 (5)
External ear pain (Ear and labyrinth disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 6 (7)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Blurred vision (Eye disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 4 (4)
Eye pain (Eye disorders) | 2 (2)
Eyelid function disorder (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 8 (11)
Dysphagia (Gastrointestinal disorders) | 8 (11)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 15 (20)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8)
Edema face (General disorders) | 1 (1)
Facial pain (General disorders) | 2 (2)
Fatigue (General disorders) | 33 (47)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Allergic reaction (Immune system disorders) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 24 (32)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 15 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 4 (5)
Dizziness (Nervous system disorders) | 5 (6)
Dysarthria (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 9 (9)
Dysphasia (Nervous system disorders) | 2 (2)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (17)
Memory impairment (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 7 (7)
Sinus pain (Nervous system disorders) | 2 (2)
Stroke (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 7 (8)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 12 (13)
Personality change (Psychiatric disorders) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (6)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT01449149/Prot_SAP_000.pdf